CLINICAL TRIAL: NCT02077712
Title: A Randomised Comparison of Two Intranasal Dexmedetomidine Doses for Ophthalmic Examination Following Failed Chloral Hydrate Sedation in Children
Brief Title: Intranasal Dexmedetomidine Sedation for Ophthalmic Examinations in Children
Acronym: DEX-EYE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Ophthalmologist, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CCPMOH2010-China4
Record Dates: First submitted 2014-02-27; First posted 2014-03-04 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Sniffs Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine 1 ug/kg (Active Comparator): 1 ug/kg of intranasal dexmedetomidine
  Interventions: Drug: intranasal dexmedetomidine
- Dexmedetomidine 2 ug/kg (Active Comparator): 2 ug/kg of intranasal dexmedetomidine
  Interventions: Drug: intranasal dexmedetomidine

INTERVENTIONS:
Drug: intranasal dexmedetomidine — 1 or 2 ug/kg of intranasal dexmedetomidine
  Other Names: Ai Bei Ning

SUMMARY:
2 ug/kg of intranasal dexmedetomidine could produce satisfactory sedation in more children for ophthalmic examinations than the sedative effect of 1ug/kg.

DETAILED DESCRIPTION:
Dexmedetomidine is an a2-adrenergic receptor agonist that provides sedation without respiratory depression.Clinical trials have demonstrated that intranasal dexmedetomidine in a dose of 1ug/kg produces satisfactory sedation in between 53% and 57% of children at anaesthetic induction. There are also reports using higher doses of intranasal dexmedetomidine. The investigators compared the sedative effect of 1ug/kg intranasal dexmedetomidine with those of 2 ug/kg for ophthalmic examinations in children aged 2 months-10 years and hypothesised that the higher dose would produce satisfactory sedation in more children at the time of anaesthetic induction.

ELIGIBILITY:
Inclusion Criteria:

* Need sedation for ophthalmic examinations
* Children who had failed chloral hydrate sedation, i.e.there was no evidence of sedation 30 min following administration.
* With informed consent from parents

Exclusion Criteria:

* Children with gastroesophageal reflux
* Children with nausea and vomiting
* Children with apnea in the past three months
* Children with recent pneumonia, exacerbation of asthma, bronchitis and upper respiratory tract infection
* Children with severe arrhythmias, heart failure and cardiac structural abnormalities
* Children with facial abnormalities, who is expected to be difficult with effective mask ventilation
* Children with severe neurological disease
* Children with moyamoya disease
* Children who is allergy to For dexmedetomidine or chloral hydrate
* Preterm children, weight <2 kg

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with successful rescue sedation | 1 day

SECONDARY OUTCOMES:
Numbers of participants with completement of ophthalmic examinations | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Xiaoliang Gan, Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ambi US, Joshi C, Ganeshnavar A, Adarsh E. Intranasal dexmedetomidine for paediatric sedation for diagnostic magnetic resonance imaging studies. Indian J Anaesth. 2012 Nov;56(6):587-8. doi: 10.4103/0019-5049.104588. No abstract available. PMID 23325950
- [Background] Ray T, Tobias JD. Dexmedetomidine for sedation during electroencephalographic analysis in children with autism, pervasive developmental disorders, and seizure disorders. J Clin Anesth. 2008 Aug;20(5):364-368. doi: 10.1016/j.jclinane.2008.03.004. PMID 18761245
- [Result] Li BL, Yuen VM, Song XR, Ye J, Ni J, Huang JX, Irwin MG. Intranasal dexmedetomidine following failed chloral hydrate sedation in children. Anaesthesia. 2014 Mar;69(3):240-4. doi: 10.1111/anae.12533. Epub 2014 Jan 21. PMID 24447296
- [Derived] Fong CY, Lim WK, Li L, Lai NM. Chloral hydrate as a sedating agent for neurodiagnostic procedures in children. Cochrane Database Syst Rev. 2021 Aug 16;8(8):CD011786. doi: 10.1002/14651858.CD011786.pub3. PMID 34397100
- [Derived] Gan X, Lin H, Chen J, Lin Z, Lin Y, Chen W. Rescue Sedation With Intranasal Dexmedetomidine for Pediatric Ophthalmic Examination After Chloral Hydrate Failure: A Randomized, Controlled Trial. Clin Ther. 2016 Jun;38(6):1522-1529. doi: 10.1016/j.clinthera.2016.04.036. Epub 2016 May 24. PMID 27229908
- See also: Homepage of Zhongshan Ophthalmic Center — http://www.gzzoc.com